CLINICAL TRIAL: NCT06054217
Title: Evaluating the Effect of Two Dosing Regimens of an Exploratory Vehicle on Meibomian Gland Dysfunction in Patients With Demodex Lid Infestation
Brief Title: Effect of an Exploratory Vehicle on Meibomian Gland Dysfunction in Patients With Demodex
Acronym: Rhea
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRS-021
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Meibomian Gland Dysfunction; Demodex Infestation of Eyelid; Blepharitis; Demodectic Blepharitis
Keywords: Demodex
MeSH Terms: conditions — Meibomian Gland Dysfunction; Blepharitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Cohort 1 (Experimental): Participants who were previously enrolled, dosed, and completed approximately 43 days of TID EV administration. Participants are crossed over to receive BID administration of EV for approximately 43 additional days.
  Interventions: Drug: Vehicle of TP-03
- Study Cohort 2 (Experimental): Participants are randomized to receive BID administration of EV for approximately 85 days.
  Interventions: Drug: Vehicle of TP-03
- Study Cohort 3 (Experimental): Participants are randomized to receive TID administration of EV for approximately 85 days
  Interventions: Drug: Vehicle of TP-03

INTERVENTIONS:
Drug: Vehicle of TP-03 — The Exploratory Vehicle is the vehicle of TP-03 (lotilaner ophthalmic solution, 0.25%)
  Other Names: Exploratory Vehicle

SUMMARY:
The purpose of this study is to evaluate and compare the effect of two dosing regimens, BID versus TID dosing, of an Exploratory Vehicle (EV) on meibomian gland dysfunction (MGD) in patients with Demodex lid infestation.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled, three-arm, investigator- and interpreter-masked study. This study is intended to compare the effect of two dosing regimens of an exploratory vehicle on meibomian gland dysfunction (MGD) in participants with Demodex lid infestation. Approximately 12 participants will be enrolled in each arm. The administration period will last for approximately 85 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Be willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol
* Meets all of the following criteria in at least one eye: have more than 10 lashes with collarettes present on the upper lid; have the presence of one or more mites with lash epilation of the upper and lower lids; have evidence of meibomian gland dysfunction; have at least mild erythema of the lower lid; have a tear breakup time of less than 10 seconds; and have intact partial to full meibomian glands in at least 33% of the total meibomian gland area of the lower lid

Key Exclusion Criteria:

* Have used lid hygiene products within 7 days of Day 1 or unwilling to forego the use of lid hygiene products during the study
* Have used systemic antihistamines within 30 days of Day 1
* Have used artificial eyelashes, eyelash extensions, or had other cosmetic eyelash or eyelid procedures within 7 days of Day 1 or be unwilling to forego their use during the study
* Contact lens wear within 7 days of Day 1 or unwilling to forego contact lens wear for the duration of the study
* Be pregnant or lactating at Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | 85 days
  TEAEs related (definitely or potentially) to treatment summarized by MedDRA preferred term.
  TEAEs related (definitely or potentially) to treatment summarized by MedDRA preferred term.

SECONDARY OUTCOMES:
Change from baseline in lower lid meibomian gland secretion score | 85 days
  For each of the 15 glands expressed, secretion characteristics will be graded via slit lamp examination on a scale of 0 to 3 (3=clear liquid secretion; 2=cloudy liquid secretion; 1=granularly opaque liquid secretion to inspissated/toothpaste consistency; and 0=no secretion).
Change from baseline in lid margin erythema. | 85 days
  Erythema of the eyelid margin will be assessed via slit lamp examination and graded on a scale of 0 (normal) to 3 (severe) for the upper and lower eyelids of each eye.
Change from baseline in tear breakup time assessed via slit lamp | 85 days
  Tear breakup time will be assessed via slit lamp examination and timed in seconds to two significant digits.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell C Shultz, MD, Principal Investigator — Shultz Chang Vision
Locations (2):
- United States (2):
  - Shultz Chang Vision, Northridge, California
  - Vita Eye Clinic, Shelby, North Carolina

IPD SHARING:
Plan to Share IPD: No